CLINICAL TRIAL: NCT03753061
Title: The Safety and Efficacy of Intracranial Thrombosis Aspiration Catheter for Recanalization in Acute Ischemic Stroke Therapy- A Prospective, Multicenter, Open Label, Blinded, Randomized Controlled, Non-inferiority Study
Brief Title: Intracranial Thrombosis Aspiration Catheter for Recanalization in Acute Ischemic Stroke Therapy (RECOVER)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Zhongrong Miao, Chief of the Department of Interventional Neurology in Beijing Tiantan Hopital, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEMO-CS1802
Record Dates: First submitted 2018-11-21; First posted 2018-11-26 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Large Vessel Occlusion; Acute Ischemic Stroke; Cerebrovascular Disorders
Keywords: Large vessel occlusion; Acute ischemic stroke; Endovascular treatment; Mechanical thrombectomy; Aspiration Catheter
MeSH Terms: conditions — Ischemic Stroke; Cerebrovascular Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspiration Catheter (Experimental): Mechanical thrombectomy with Aspiration Catheter.
  Interventions: Device: Aspiration Catheter
- Stent Retriever (Solitaire FR) (Active Comparator): Mechanical thrombectomy with Solitaire FR.
  Interventions: Device: Solitaire FR

INTERVENTIONS:
Device: Aspiration Catheter — Patients will be treated for mechanical recanalization with Aspiration Catheter within 8 hours after stroke onset plus standard medical management.
  Arms: Aspiration Catheter
Device: Solitaire FR — Patients will be treated for mechanical recanalization with Solitaire FR within 8 hours after stroke onset plus standard medical management.
  Arms: Stent Retriever (Solitaire FR)

SUMMARY:
This study is a prospective, multi-center, open-label, end-point blinded, randomized, parallel positive control, non-inferiority clinical trial, with a purpose to evaluate the safety and efficacy of Hemo Jirui intracranial thrombus aspiration catheter system for endovascular treatment of acute ischemic stroke by comparison with stent retriever (Solitaire FR). The trial is anticipated to last from November 2018 to May 2019, with 204 subjects recruited from 15-20 clinical trial centers in China.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, open-label, end-point blinded, parallel positive controlled, non-inferiority clinical trial. Patients with acute ischemic stroke (AIS) who meet inclusion criteria would be enrolled in this study. Led by Beijing Tiantan Hospital affiliated to Capital Medical University, this study is planned to be carried out in 15-20 clinical trial institutions in China. There will be 102 patients enrolled in each group. Patients in the experimental group will be treated with the intracranial thrombus aspiration catheter, product of Hemo Jirui. Patients in the control group will be treated with stent retriever (Solitaire FR).

In this trial, relevant examinations of safety and efficacy assessments were performed immediately after the procedure, at 24 hours, 7 days, 30 days, and 90 days. Primary efficacy endpoint will be the immediate recanalization rate (mTICI 2b-3) of target vessel after the procedure. Secondary efficacy endpoints will include: (1) Proportion of functional independence (mRS 0-2) at 90 days; (2) ordinal shift analysis of mRS at 90 days; (3) immediate recanalization rate (mTICI 2b-3) of the first pass of thrombectomy device; (4) immediate recanalization rate (mTICI 2b-3) of the last pass of thrombectomy device; (5)procedure time (randomization to recanalization); (6) Change in NIHSS score at 24hours; (7) Change in NIHSS score at 7 days or discharge (whichever comes first); (8) mTICI grading of target vessel revealed by CTA or MRA at 22-36 hours; (9) The extent of anterior circulation infarction at 22-36 hours, as measured by ASPECTS on CT or MRI. Safety endpoints will include: (1) All-cause mortality at 90 days; (2) stroke-related mortality at 90 days; (3) stroke recurrence rate within 90 days; (4) any type of intracranial hemorrhagic transformation within 22-36 hours, including parenchymal, subarachnoid or ventricular hemorrhage; (5) symptomatic intracranial hemorrhage (sICH) within 22-36 hours, as confirmed by any intracranial hemorrhage on CT or MRI associated with ≥ 4 points of worsening on NIHSS or even contributing to death; (5) procedural complications or serious adverse events procedural complications or serious adverse events (SAEs) within 90 days.

The trial is anticipated to last from November 2018 to May 2019, all the related investigative organization and individuals will obey the Declaration of Helsinki and Chinese Good Clinical Practice standard. The trial has been approved by Institutional Review Board (IRB) and Ethics Committee(EC) in Being Tiantan hospital, Capital Medical University.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Symptoms and signs in accordance with anterior circulation ischemia and large vessel occlusion (ICA, MCA-M1 or M2) confirmed by CTA/MRA/DSA.
3. Pre-stroke Modified Rankin Scale（mRS）0-1.
4. NIHSS score ≥ 6 points at time of randomization.
5. The patients should receive endovascular treatment within 8 hours of estimated time of large vessel occlusion (LVO) onset, and have an ASPECTS ≥ 6 points on non-enhanced CT.
6. If intravenous thrombolysis with tPA (IVT) is considered as part of standard medical management, IVT should be started within 4.5 hours of estimated time of LVO. Furthermore, in AIS patients with an unknown time of onset, IVT guided by a mismatch between DWI and FLAIR in the region of ischemia is also recommended.
7. Written informed consent obtained from patient or patient's legally authorized representative.

Exclusion Criteria:

1. Acute posterior circulation cerebral infarction comfirmed by CT or MRI.
2. Any type of cerebral hemorrhage (only microbleeds are allowed) on neuroimaging.
3. Large (more than one-third of the MCA) regions of clear hypodensity on the baseline CT scan or ASPECTS < 7 points or significant mass effect with midline shift.
4. Proven occlusion of the common carotid artery.
5. Known or suspected chronic occlusion of target vessel.
6. Known life threatening allergy (more than rash) to iodinated contrast agent.
7. Arterial tortuosity and other problems that would prevent the device from reaching the target vessel.
8. Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency.
9. Baseline platelet count < 50000/µL.
10. Severe heart, liver or kidney failure and other serious or terminal illness.
11. Major surgery within the past 2 weeks
12. Haemorrhage of the gastrointestinal or urinary tract within the past 3 weeks.
13. Baseline blood glucose < 2.7 or > 22.2 mmol/L.
14. Baseline blood pressure > 185/110 mmHg, or aggressive treatment (intravenous medication) necessary to reduce blood pressure to these limits
15. Pregnant or lactating or positive pregnancy test on admission.
16. Dementia or psychiatric disease that would confound the neurological or functional evaluations.
17. Life expectancy less than 1 year.
18. Current participation in another drug or device research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2018-11-22 (Actual); Primary Completion 2020-03-20 (Estimated); Study Completion 2020-03-20 (Estimated)

PRIMARY OUTCOMES:
Instant recanalization rate (mTICI 2b-3) of target vessel after the procedure | immediate

SECONDARY OUTCOMES:
Proportion of functional independence (mRS 0-2) at 90 days | 90 days
Ordinal shift analysis of mRS at 90 days | 90 days
Instant recanalization rate (mTICI 2b-3) after the first thrombectomy | immediate
Instant recanalization rate (mTICI 2b-3) after the last thrombectomy | immediate
Procedure time (randomization to recanalization) | procedure
Change in NIHSS score at 24±2 hours | 24 hours
Change in NIHSS score at 7±1 days or discharge (whichever comes first) | 7 days
mTICI grading of target vessel revealed by CTA or MRA at 22-36 hours | 22-36 hours
The extent of anterior circulation infarction at 22-36 hours, as measured by ASPECTS on CT or MRI | 22-36 hours

CONTACTS AND LOCATIONS:
Locations (23):
- China (23):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Luhe Hospital Medical University, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Tangshan People's Hospital, Tangshan, Hebei
  - Luoyang Central Hospital, Luoyang, Henan
  - Henan Province People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhengzhou Central Hospital, Zhengzhou, Henan
  - Taihe Hospital, Shiyan, Hubei
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Baotou Central Hospital, Baotou, Neimenggu
  - Tangdu Hospital, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Qingdao Central Hospital, Qingdao, Shandong
  - Weihai Central Hospital, Weihai, Shandong
  - Yantaishan Hospital, Yantai, Shandong
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality